CLINICAL TRIAL: NCT06081868
Title: A Randomized Clinical Trial on the Effectiveness of Oral Health Preventive Programmes in School Children in Uganda
Brief Title: RCT on Effectiveness of Oral Health Preventive Programmes in School Children in Uganda
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was put in hold due to COVID Pandemic and we are still in discussion when to to restart
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Bernzmk20072023
Record Dates: First submitted 2023-09-06; First posted 2023-10-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Dental Caries; Dental Plaque; Dental Diseases; Dental Caries in Children; Oral Disease; Oral Manifestations
Keywords: Oral health; Prevention programme; Randomized controlled trial; Sustainable healthy habits; Uganda
MeSH Terms: conditions — Dental Caries; Dental Plaque; Stomatognathic Diseases; Mouth Diseases; Oral Manifestations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toothbrush/toothpaste/fluoride varnish (Experimental): Children will be instructed to use toothbrush/toothpaste/fluoride varnish.
  Interventions: Behavioral: Use of toothbrush/toothpaste/fluoride varnish
- Education on nutrition/oral hygiene (Experimental): Children receive individual education on nutrition/oral hygiene.
  Interventions: Behavioral: Education on nutrition/oral hygiene

INTERVENTIONS:
Behavioral: Use of toothbrush/toothpaste/fluoride varnish — Children receive information about the use of toothbrush/toothpaste/fluoride varnish.
  Arms: Toothbrush/toothpaste/fluoride varnish
Behavioral: Education on nutrition/oral hygiene — Children receive education on nutrition/oral hygiene.
  Arms: Education on nutrition/oral hygiene

SUMMARY:
Dental caries represents a challenge for Oral Health Services in several African Countries, like Uganda. Few studies have been reported the burden of oral health, its prevention and non-operative treatment among school children in African countries.

Aim: To assess the prevalence and risk factors of dental caries and the effectiveness of strategies to prevent and treat dental caries using a non-operative approach among children in Gulu Municipality, Uganda.

Methods: The proposal RCT is structured in three phases: 1. A descriptive cross-sectional survey to collect oral data among 610 school children selected using a multistage cluster sampling; 2. A randomized unblinded two-arm trial to assess the difference in the treatment/prevention of dental caries using non-operative means among school children in the Ugandian Gulu municipality; and 3. A comparison of oral health conditions between a group of children who will be given dental cleaning tools and followed up over time versus a control group.

The oral health status of the participants will be assessed according to WHO and ICDAS guidelines. Stata 14.0. will be used for analysis; descriptive statistics will be carried out to analyze continuous and categorical variables and chi-square test as well as independent tests for bivariate analysis and modified poisson regression. In addition, the factors associated with dental caries will be determined by linear regression models using a statistical significance level of 5% (α = 0.05).

Discussion: This trial will be the first trial conducted in Uganda assessing a school-based caries prevention programme using the WHO and ICDAS standardized international guidelines. The findings obtained will increase knowledge on oral health in Uganda school children and the effectiveness of community-based caries prevention programme in this population.

DETAILED DESCRIPTION:
Study design

This randomized controlled clinical study will be developed in three parts: 1.) An epidemiological survey; a descriptive cross-sectional study to be conducted in Gulu Municipality to collect data on the oral health of school children to assess caries prevalence and associated factors. 2.) A field trial; an individually randomized, unblinded, two-armed trial of toothbrush/toothpaste/fluoride varnish versus education on nutrition/oral hygiene to assess the difference in treatment/prevention of dental caries. 3.) A comparison of oral health conditions among a group of children who were provided with dental cleaning tools and who were followed up and monitored over time versus a control group.

Study setting and location

The study will be conducted in Gulu Municipality, Gulu District, in Northern Uganda. The municipality has four sub-counties, each consisting of four parishes, with a total population of 177'400 according to the Uganda Bureau of Statistics (UBOS), 2020 projection [Uganda Bureau of Statistics in Uganda. April 2019 Population Projections by Subcounty and Sex (2015-2030), in Population & Censuses. 2019]. It is the largest urban center in Acholi sub-region. There are three hospitals offering oral health services in Gulu Municipality: Gulu referral hospital, St. Mary's Hospital, Lacor and Gulu independent hospital. Primary schools in Gulu Municipality will be used as study areas. The list of primary schools in the Municipality will be obtained from the District Education Officer (DEO). An ethical approval from the Ministry of Health and consents from parents of the school children will be required.

Study population

The study will be conducted among school children in Gulu Municipality for 24 months, starting in September 2024. The inclusion criteria will be: enrollment in one of primary schools in Gulu Municipality, age between 5 and 17 years, staying in the area for at least six months and parent/guardian's willingness to give consent. Exclusion criteria will be: school children who refuse to participate in the research and/or parents who refuse their children's participation and children with chronic diseases or systemic conditions that require differential care and follow-up.

Data collection

A modified World Health Organization (WHO) questionnaire on children oral health [Oral health surveys: basic methods. 2013: World Health Organization.] will be used for each participant to identify factors such as socioeconomic status, dietary habits, oral health habits, and dental attendance associated with oral health data.

The dental examinations will be performed by five trained and calibrated dentists. These will receive an intensive two-day training session of at least 72 hours together with a demonstration on images depicting carious lesions of varying severity in order to learn how to assess them through the International Caries Detection and Assessment System [Dikmen, B., ICDAS II criteria (International Caries Detection and Assessment System). Journal of Istanbul University Faculty of Dentistry, 2015;49(3):63.].

A benchmark examiner will calibrate the examiners' practice on caries detection to ensure accurate and correct application of the research procedures. The first ten enrolled participants will be used for calibration exercise. The unweighted kappa statistic will be used to assess the inter-examiner and intra-examiner agreement. The dental examination will be carried out using a mirror and a probe, under appropriate artificial light and after cleaning the teeth with cotton rolls to remove food debris and dental plaque. Oral health status will be evaluated according to the method and criteria recommended by the WHO [Oral health surveys: basic methods. 2013: World Health Organization.], including the ICDAS [Dikmen, B., ICDAS II criteria (International Caries Detection and Assessment System). Journal of Istanbul University Faculty of Dentistry, 2015;49(3):63.].

The following data will be collected after obtaining consent and enrolment:

* Date of enrolment
* Date and time of consent
* Participant identifiers
* Socio-economic and demographic information
* Status of the oral health

Follow up visits:

* All participants will be re-assessed clinically every three months after enrolment until the 24th month to evaluate oral health status. A symptom checklist, targeted dental examinations and a record of the findings and treatments administered will be performed at each visit.
* All costs related to the health care of the project participants will be recorded, starting from enrolment and for the duration of follow-up. The costs will also include those for any hospitalisation related to dental caries and those arising from the use of other health care resources, including the costs of materials used for each visit.

Project variables

The first part of this project is an epidemiological survey in which the prevalence of dental caries will be the primary outcome. The outcome will be calculated by determining the percentage of participants diagnosed with dental caries, while the secondary outcome will be the extent of other oral diseases. The mean values of carious teeth/surfaces, missing teeth/surfaces, filled teeth/surfaces and mean DMFT/S will be calculated. A questionnaire will be used to investigate the relationships between the prevalence of dental caries and other variables such as sex, demographic information, school, age, hygiene habits (brushing frequency), maternal education, dietary habits (frequency of mealtimes, frequency of sugar intake, sugar intake between meals, soft drink consumption between meals).

The second phase of the project is a field trial in which the outcome variable will be the presence of dental caries after the intervention. Secondary outcomes will include resolution of dental caries symptoms, cost of interventions performed.

A full study protocol will be published in a peer-reviewed journal in a timely manner and will be included here afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in one of primary schools in Gulu Municipality
* Age between 5 and 17 years
* Staying in the area for at least six months
* Parent/guardian's willingness to give consent
* Written informed consent by participant and/or parents

Exclusion Criteria:

* School children who refuse to participate in the research
* Parents who refuse their children's participation
* Children with chronic diseases or systemic conditions that require differential care and follow-up

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 610 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dental caries | Baseline
  The outcome will be calculated by determining the percentage of participants diagnosed with dental caries.
Prevalence of dental caries | 12 months
  The outcome will be calculated by determining the percentage of participants diagnosed with dental caries.
Prevalence of dental caries | 24 months
  The outcome will be calculated by determining the percentage of participants diagnosed with dental caries.
Mean of dental caries | Baseline
  The mean values of carious teeth/surfaces, missing teeth/surfaces, filled teeth/surfaces and mean DMFT/S will be calculated.
Mean of dental caries | 12 months
  The mean values of carious teeth/surfaces, missing teeth/surfaces, filled teeth/surfaces and mean DMFT/S will be calculated.
Mean of dental caries | 24 months
  The mean values of carious teeth/surfaces, missing teeth/surfaces, filled teeth/surfaces and mean DMFT/S will be calculated.
Presence of dental caries after the intervention | Baseline
  The outcome will be calculated by determining the percentage of participants diagnosed with dental caries. The mean values of carious teeth/surfaces, missing teeth/surfaces, filled teeth/surfaces and mean DMFT/S will be calculated.
Presence of dental caries after the intervention | 12 months
  The outcome will be calculated by determining the percentage of participants diagnosed with dental caries. The mean values of carious teeth/surfaces, missing teeth/surfaces, filled teeth/surfaces and mean DMFT/S will be calculated.
Presence of dental caries after the intervention | 24 months
  The outcome will be calculated by determining the percentage of participants diagnosed with dental caries. The mean values of carious teeth/surfaces, missing teeth/surfaces, filled teeth/surfaces and mean DMFT/S will be calculated.

SECONDARY OUTCOMES:
Extent of other oral diseases | Baseline
  The presence of other oral diseases and manifestations is documented upon examination.
Extent of other oral diseases | 12 months
  The presence of other oral diseases and manifestations is documented upon examination.
Extent of other oral diseases | 24 months
  The presence of other oral diseases and manifestations is documented upon examination.
Cost of clinical interventions | Baseline
  The costs incurred for the measures implemented in each case are identified and investigated.
Cost of clinical interventions | 12 months
  The costs incurred for the measures implemented in each case are identified and investigated.
Cost of clinical interventions | 24 months
  The costs incurred for the measures implemented in each case are identified and investigated.
Identification of dental caries symptoms | Baseline
  Sign or symptoms for caries will be investigated using ICDAS International Caries Detection and Assessment System (Scale from 0 healthy (best score) to 6 pulp involvement (worst score))
Identification of dental caries symptoms | 12 months
  Sign or symptoms for caries will be investigated using ICDAS International Caries Detection and Assessment System (Scale from 0 healthy (best score) to 6 pulp involvement (worst score))
Identification of dental caries symptoms | 24 months
  Sign or symptoms for caries will be investigated using ICDAS International Caries Detection and Assessment System (Scale from 0 healthy (best score) to 6 pulp involvement (worst score))

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Wolf, DDS,MA,Prof, Principal Investigator — University of Bern, Switzerland; Guglielmo Campus, DDS,PhD,Prof, Principal Investigator — Uniersity of Bern, Switzerland; Obaida El-Modalal, DDS, Study Director — University of Bern, Switzerland; Maria-Grazia Cagetti, DDS,PhD,Prof, Study Director — University of Milan, Italy; Hannington Baliddawa, DDS, Dr., Study Director — Uganda Dental Association, Uganda; Dominique Corti, MD, Dr., Study Director — Corti Foundation, Uganda; Friedrich Herbst, Study Director — Academy of Dentistry International, USA; Philippe Rusca, DDS, Dr., Study Director — University of Bern, Switzerland
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No